CLINICAL TRIAL: NCT02584985
Title: A Multicentric Randomised Trial to Evaluate Efficacy, Morbidity and Functional Outcome of Endoscopic TranAnal Proctectomy Versus Standard Transabdominal Laparoscopic Proctectomy for Low Lying Rectal Cancer (ETAP-GRECCAR 11)
Brief Title: Evaluate Efficacy, Morbidity and Functional Outcome of Endoscopic TranAnal Proctectomy vs Standard Transabdominal Laparoscopic Proctectomy for Rectal Cancer
Acronym: ETAP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETAP-GRECCAR 11-IPC 2015-005
Record Dates: First submitted 2015-10-15; First posted 2015-10-23 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETAP : Endoscopic Transanal Proctectomy (Other): 1. Primary transanal approach :
     Careful positioning in Lithtomy, dilatation and anal exposure with standard retractor. Mucosa incision and internal sphincter dissection according to tumor extension. Primary conventional dissection up to circumferential exposure of fascia recti. Secondary implantation of transanal endoscopic device Begin mesorectal endoscopic dissection postero-anteriorly, then laterally with nerve-sparing dissection. Level assessment of posterior dissection (vertical segment). End with peritoneal opening anteriorly (Douglas).
  2. Secondary transabdominal approach :
  Type of laparoscopic approach multiport or singleport. Level of arterial section, extension of colonic mobilization, site for specimen extraction (transanal / transabdominal), type of colonic reconstruction.
  Interventions: Procedure: ETAP
- Standard Transabdominal Laparoscopic proctectomy (Other): Primary transanal conventional dissection (sphincter preservation assessment) or not, type of laparoscopic approach multiport or singleport, level of arterial section, extension of colonic mobilization, conditions of mesorectal excision and nerve preservation, site for specimen extraction (transanal / transabdominal) and type of colonic reconstruction.
  Interventions: Procedure: Standard Transabdominal Laparoscopic Proctectomy

INTERVENTIONS:
Procedure: ETAP — Primary transanal endoscopic approach, secondary transabdominal laparoscopic approach
  Arms: ETAP : Endoscopic Transanal Proctectomy
Procedure: Standard Transabdominal Laparoscopic Proctectomy — Primary transabdominal laparoscopic approach
  Arms: Standard Transabdominal Laparoscopic proctectomy

SUMMARY:
Standard surgical treatment of mid and low rectal cancer is total mesorectal excision (TME). Originally performed by open surgery, TME demonstrated improved local control and reduced urogenital morbidity. Laparoscopic approach has been validated by several randomised controlled trials: laparoscopic approach offers to the patient a better post-operative recovery, a lower risk of wound hernia and comparable oncological results. However, the risk of conversion to open procedure remains significant.

Endoscopic Transanal Proctectomy allows retrograd mesorectal excision, performing the whole pelvic dissection via a specific-moderate cost device. The procedure is then completed by a briefer transabdominal laparoscopic step to mobilise the colon and perform inferior mesenteric vessels ligation, prior to low coloanal anastomosis. The originality of this approach is to perform a surgical dissection via an extra peritoneal route, without peritoneal and abdominal wound trauma. This focuses on new technical improvement in the area of mini-invasive pelviabdominal surgery using natural orifice as surgical access. This approach offer closer and better exposure of pelvic dissection plane and could improve oncological quality and pelvic nerve preservation. It could be profitable to postoperative patient outcome. However rates and type of cancer-recurrences as well as functional results have to be assessed in a controlled study. This technique has shown to be feasible and reproducible through early clinical series. Conversion rates appear to be lower than published rates of laparoscopic approach, markedly inferior to 10%. Compiled rates of morbidity (27.8%), R1 resection* (6%), mesorectum macroscopic integrity (100%) appear to be comparable to laparoscopic approach results. However functional results as well as urologic morbidity have to be evaluated in comparative studies. In a preliminary retrospective comparative (n=72) we founded comparable oncological quality criteria (R1 resection 5.9% vs 10.5% p 0.74, Grade 3 mesorectal integrity 57.5 vs 56.2 p 0.99), lower conversion rate to open procedure (2.9% vs 23.6% p 0.011), shorter in-hospital stay (8 vs 9 days p 0.038). Comparable morbidity rates (Dindo 1-4 27% vs 34% p 0.52) and functional results (Kirwan 1/2 80.3% vs 80.6% p 0.94) were also founded. These data need to be confirmed. To this date, Endoscopic Transanal Proctectomy has been evaluated through preliminary studies including several short series demonstrating the feasibility of the technique and showing low morbidity. For some authors the benefit of transanal approach is significant in difficult cases such as male patient and narrow pelvis. Very recently, two non randomised comparative studies were published with conclusions close to those in our study.

Investigators propose, with the support of the GRECCAR group, to conduct a national, multicenter, open-label randomized study based on oncological non-inferiority (R1 resection rate) for the main objective, comparing Endoscopic Transanal Proctectomy to Standard Transabdominal Laparoscopic Proctectomy, for low lying rectal cancer requiring manual colo-anal anastomosis. There is a clear expected benefit expected for the patients through the ETAP procedure in term of post operative short term outcome, risk of conversion to open procedure, risk of wound hernia.This trial could also show significant advantages in terms of quality of dissection, quality of the specimen, quality of nerve preservation.

DETAILED DESCRIPTION:
The main objective of study is to assess if R1 resection rate of Endoscopic Transanal Proctectomy (ETAP) is not meaningfully inferior to Standard Laparoscopic TME for low lying rectal cancer requiring manual colo-anal anastomosis. The secondary objective will evaluate conversion rate, mini invasive level of abdominal approach postoperative morbidity, In hospital length of stay, Mesorectum macroscopic assessment, Functional urologic and sexual results, Fecal Continency, global QoL, stoma-free survival, disease-free survival at 3 years. Patients with non metastatic rectal adenocarcinoma requiring coloanal anastomosis will be considered for the study. Based on the non-inferiority hypothesis, the population estimated in this study at 226 patients, 113 for each arm. Inclusion period will be 3 years, the study will be running for 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Non metastatic stadified T3 rectal adenocarcinoma allowing sphincter-sparing procedure
* Tumor location or local condition justifying manual coloanal anastomosis
* Age >18 years
* Patient eligible for surgery
* Written informed consent
* Affiliation to Social Security System

Exclusion Criteria:

* Tumor stadified T4 with en-bloc resection
* Possible mechanical trans-sutural anastomosis
* Distant metastasis at diagnosis
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule
* Patients deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
R1 resection rate | from surgery up to 3 years
  R1 resection rate defined as circumferential resection margin (CRM) ≤ 1 mm, distal or positive margin (and the complete rectal resection meso levels (grade III) as classified by Quirke).

SECONDARY OUTCOMES:
Failure rate (conversion to open) | During surgery
Disease-free survival at 3 years | 3 years from surgery

CONTACTS AND LOCATIONS:
Overall Officials: LELONG Bernard, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

REFERENCES:
- [Derived] Lelong B, de Chaisemartin C, Meillat H, Cournier S, Boher JM, Genre D, Karoui M, Tuech JJ, Delpero JR; French Research Group of Rectal Cancer Surgery (GRECCAR). A multicentre randomised controlled trial to evaluate the efficacy, morbidity and functional outcome of endoscopic transanal proctectomy versus laparoscopic proctectomy for low-lying rectal cancer (ETAP-GRECCAR 11 TRIAL): rationale and design. BMC Cancer. 2017 Apr 11;17(1):253. doi: 10.1186/s12885-017-3200-1. PMID 28399840
- See also: Institut PAOLI-CALMETTES — http://www.institutpaolicalmettes.fr